CLINICAL TRIAL: NCT05110040
Title: A Multi-model Image of Immunosuppressive Agents in Thyroid Associated Ophthalmopathy.
Brief Title: Multi-model Image of Immunosuppressive Agents in TAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, Dan Liang, PhD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAOIMTIMAGE
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Thyroid Associated Ophthalmopathy
Keywords: Thyroid Associated Ophthalmopathy; Immunosuppressive agents; multi-modal image; function assessment
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Immunosuppressive Agents

STUDY DESIGN:
Intervention Model Description: participants diagnosed of TAO administrated with immunosuppressive agents
Masking Description: Assessors who calculate the changes of the images are masked of the diagnosis and treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immunosuppressive agents (Experimental): patients recruited will be treated with one or／and two immnuosuppressive agents
  Interventions: Drug: immunosuppressive agent

INTERVENTIONS:
Drug: immunosuppressive agent — patients with TAO recruited in this study will administrated with immunosuppressive agent per day
  Other Names: immunosuppressive regulator

SUMMARY:
This study aims to evaluate the efficacy of immunosuppressive agents treating Thyroid Associated Ophthalmopathy by multi-model image.

DETAILED DESCRIPTION:
Thyroid Associated Ophthalmopathy is one of autoimmune orbital diseases characterized by enlargement of the extraocular muscles and increase in fatty or/and orbit connective tissue volume affecting the appearance and visual function of the eyes. TAO can be classified into active phase and inactive phase according to the activity score and wait-and-see or surgery are widely chosen for patients in inactive phase. A great number of patients in inactive phase becoming refractory and reoccurring.

Until now, the improvement of TAO is still be measured subjectively with low reliability and less accuracy. Multi-modal image is a new method to assess both the appearance and visual function of TAO and some of the indexes can be regarded as more apparent and stable in assessing the efficacy and prognosis of TAO.

This perspective cohort study aims to evaluate the efficacy of immunosuppressive agents in TAO by multi-model image and function assessments.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 18-70 years old
* Diagnosed with TAO.

Exclusion Criteria:

* Contraindications to immunosuppressive agents.
* Patients with HIV, Hepatitis B or C, Tuberculosis or other active significant infection.
* Patients with severe chronic diseases in heart, lung, kidney and liver, which make it not tolerant to immunosuppressive agents.
* Patients have contraindications of MRI(metal pacemaker, fake teeth, foreign body and other materials which will disturb the examination).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
change of macular sensibility | At 6 months
  the same investigator uses the same instrument to assess the macular sensibility. The better change of macular sensibility means the better outcome.

SECONDARY OUTCOMES:
change of extraocular muscle volume and orbital fat volume by MRI | at month 6
  A 3D MRI reconstructive model will be established and the volume of extraocular muscle and orbital fat will be calculated by the same advanced programmer who is blinded of the pre- or post- treatment images order. The higher the value changes, the better the outcome is.
change of proptosis | at month 6
  proptosis will be measured by the same investigator using the same Hertel instrument
change of QoL | at month 6
  the score of quality of life will be assessed by the same investigator using GO-QoL. The higher change of quality of life means the better outcome.
change of eyelid aperture and lid lag | at month 6
  the values will be measured by the same investigator using the same millimeter ruler and the higher change of eyelid aperture and lid lag means the better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No